CLINICAL TRIAL: NCT04171284
Title: A Multicenter Randomized Double-blinded Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of SCT-I10A or Placebo Plus Docetaxel in Treating Advanced Squamous Non-small Cell Lung Cancer
Brief Title: SCT-I10A or Placebo Plus Docetaxel With Previously Treated Squamous Cell Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategy adjustments, independent of the safety and efficacy of the trial medication
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCT-I10A-D301
Record Dates: First submitted 2019-11-12; First posted 2019-11-20 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Squamous-cell Non-Small-cell Lung Cancer
Keywords: Non-small cell lung cancer; Squamous cell carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell | interventions — Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SCT-I10A plus Docetaxel (Experimental): SCT-I10A 200mg, I.V., Q3W; Docetaxel 70-75 mg per square meters of body surface area,I.V., Q3W. Maximum of 6 cycles
  Interventions: Drug: SCT-I10; Drug: Docetaxel
- Placebo puls docetaxel (Active Comparator): Placebo 200mg, I.V., Q3W; Docetaxel 70-75 mg per square meters of body surface area,I.V., Q3W Maximum of 6 cycles
  Interventions: Drug: Docetaxel; Drug: Placebo
- Maintenance therapy of SCT-I10A (Experimental): Subjects complete 2-6 cycles of combined therapies, when the evaluation result is CR, PR or SD (RECIST 1.1), the subjects will enter maintain therapy: SCT-I10A 200mg, I.V., Q3W, till progression, loss to follow-up, new antineoplastic therapy or intolerable toxicity.
  Interventions: Drug: SCT-I10
- Maintenance therapy of Placebo (Placebo Comparator): Subjects complete 2-6 cycles of combined therapies, when the evaluation result is CR, PR or SD (RECIST 1.1), the subjects will enter maintain therapy: Placebo 200mg, I.V., Q3W, till progression, loss to follow-up, new antineoplastic therapy or intolerable toxicity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCT-I10 — 200 mg, Q3W, maximum treatment up to six cycles
  Other Names: human PD-1 monoclonal antibody
  Arms: Maintenance therapy of SCT-I10A; SCT-I10A plus Docetaxel
Drug: Docetaxel — 70-75mg per square meters of body surface area, Q3W, maximum treatment up to six cycles
  Arms: Placebo puls docetaxel; SCT-I10A plus Docetaxel
Drug: Placebo — 200 mg, Q3W, maximum treatment up to six cycles
  Arms: Maintenance therapy of Placebo; Placebo puls docetaxel

SUMMARY:
This is a phase 3 double-blinded randomized multicenter clinical trial of SCT-I10A or placebo plus docetaxel with previously treated squamous cell non-small cell lung cancer patients. The main endpoint is to compare the overall survival (OS) of these two regimens above.

DETAILED DESCRIPTION:
In 2015, there were near 787,000 patients diagnosed with lung cancer in China. And in the very same year, 631,000 lung cancer patients died of the disease. Lung cancer still causes most cancer related death in here. Approximately 85% of lung cancer is non-small cell lung cancer (NSCLC) compared with small cell lung cancer (~15%) pathologically. NSCLC include squamous cell NSCLC, adenocarcinoma and large cell carcinoma. Although there are therapies developed to treat the condition, patients with advanced squamous-cell (NSCLC) who have disease progression during or after first-line chemotherapy have limited treatment options in China. Hence, we developed a fully human IgG4 programmed death 1 (PD-1) immune-checkpoint-inhibitor monoclonal antibody (SCT-I10A) which inhibits the interaction between PD-1 and its ligands results in the reactivation of active T cell and finally leads to caner immunotherapy. We are now carrying out a phase 3 clinical trial to determine whether SCT-I10A plus docetaxel surpass docetaxel monotherapy with previously treated squamous-cell NSCLC patients. As designed in the protocol, 360 eligible subjects would be randomized into two arms in a ratio of 2:1. 240 subjects would be treated with SCT-I10A plus docetaxel in the experimental arm while 120 subjects would be treated with placebo plus docetaxel in the active comparator arm. Both of these arms will be treated with maintenance therapy after planed treatments. Our primary endpoint is overall survival, secondary endpoints are PFS, OSR, ORR, DOR, DCR and other efficacy and safety index.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be voluntarily sign the written informed consent.
2. Histologically or cytologically confirmed diagnosis of locally advanced or metastatic squamous NSCLC. Or recurrent squamous NSCLC according UICC/AJCC 8th edition.
3. At least one measurable tumor lesion per RECIST 1.1 criteria. A lesion previously irradiated could be considered as a target lesion only in the condition that progression occurred at the time of 3 months after the end of radiotherapy.
4. Previously treated with one platinum based regimen (including platinum and endostar regimen) and progression occur during or after treatment or unbearable treatment related adverse events.
5. Progression after EGFR-TKIs in patients with driver gene mutation.
6. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.

Exclusion Criteria:

1. Patient who is allergic to recombinant humanized PD-1 monoclonal antibody or the components of the drug.
2. Patient who is allergic to taxane.
3. Previously treated with any of the antibodies targeted on PD-1, PD-L1, PD-2, CD137, CTLA-4, T cell, co-stimulation or drugs targeted on the checkpoint signal pathway.
4. Previously treated with docetaxel.
5. The histopathological subtype is not squamous cell non-small cell lung cancer, or squamous cell < 90% in a mixed carcinoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to approximately 3 years
  OS is the time from the date of randomization to death due to any cause.

SECONDARY OUTCOMES:
PFS | Up to approximately 3 years
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
OSR of 6 months, 12 months and 18 moths | Each subject that randomized will be followed up for 18 months to measure the OSR.
  overall survival rate from the date of randomization till the 6 months,12 months and 18 months
ORR | Up to approximately 3 years
  ORR is the proportion of subjects with CR or PR based on RECIST v1.1.
DOR | Up to approximately 3 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
DCR | Up to approximately 3 years
  DCR is defined as the proportion of subjects with CR, PR, or SD based on RECIST v1.1.
The concentration of anti-SCT-I10A antibodies in the serum of subjects | Up to approximately 3 years
  The concentration of anti-SCT-I10A antibodies in the serum of subjects during or after the study treatments will be measured, its level could indicate the immunogenicity of SCT-I10A.
The expression level of PD-L1 of subjects' specimens | Up to approximately 3 years
  The expression level of PD-L1 of the subjects would be measure by immunohistochemical detection. The results would be used to analyze the correlation of PD-L1 level and outcomes including primary and secondary endpoints including OS, PFS, OSR, ORR, DOR and DCR.
Cancer-specific quality of life of the regimens treated subjects | Up to approximately 3 years
  European Organisation for Research and Treatment of Cancer (EORTC) cancer-specific quality of life questionnaire (EORTC QLQ-C30) will be applied in all subjects to collect the score of 30 items of subjects before and after study treatments. For the items from one to twenty-eight, the minimum and maximum scores are 28 and 112 respectively and the higher score means a worse outcome. For the items from twenty-nine to thirty, the minimum and maximum raw scores are 2 and 14 respectively and the higher score means a better outcome. Further analysis could be done based on the calculation.
Lung cancer-specific quality of life of the regimens treated subjects | Up to approximately 3 years
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13) will be applied in all subjects to collect the score of 13 specific typical symptoms of lung cancer patients before and after study treatments. The minimum and maximum raw scores are 12 and 52 respectively, the higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Han Baohui, M.D., Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han B, Wu L, Yang R, Wu H, Li W, Yu Y, Zhang M, Sun H, Chu T, Zhong F, Fang Y, Wu R, Bian T, Guo X, Sun M, Zhang Y, Liu L, Liu X, Pan Y, Jiang O, Wei Z, Lin H, Guo W, Fang J, Wang J, Ding C, Hu Y, Ye F, Zhuang W, Ye S, Wang L, Huang Z, Liu C, Yang L, Wang J, Xie L. Efficacy and safety of finotonlimab plus docetaxel vs. docetaxel in previously treated advanced squamous cell non-small-cell lung cancer: a randomized, double-blinded, phase III trial. Transl Lung Cancer Res. 2025 Apr 30;14(4):1231-1241. doi: 10.21037/tlcr-24-1042. Epub 2025 Apr 16. PMID 40386729